CLINICAL TRIAL: NCT06473558
Title: Identification of Depressive and Anxiety Symptoms Among a Sample of Emergency Department Patients Using Artificial Intelligence (AI) Technology
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY20240008
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Artificial Intelligence (AI)
Keywords: Depression; Anxiety; Emergency Department
MeSH Terms: conditions — Depression; Anxiety Disorders; Emergencies | interventions — Biometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Participants seen at University Hospitals Cleveland Medical Center Emergency Department (Experimental): Eligible patients must present with non-emergent concerns of Emergency Severity Index (ESI) level 3, 4, or 5. Patients will complete assessments and questionnaires and end with being recorded reading a story to capture facial expressions and audio cues.
  Interventions: Device: Biometrics (or AI Biomaker)

INTERVENTIONS:
Device: Biometrics (or AI Biomaker) — Patients will be asked to read a story and their facial expressions and audio cues will be recorded.

SUMMARY:
Behavioral health problems, such as depression and anxiety, are common yet often are not identified by emergency department doctors and nurses. These mental health conditions can be due to medical issues or can worsen medical problems. One way investigators hope to do a better job of learning about mental health is by training Artificial Intelligence (AI) software to detect anxiety and depression by analyzing facial expression and tone of voice.

Participants are invited to participate in a study which may help improve emergency department care. An audio and video recording of the participant's responses to some simple, non-psychological questions will be analyzed by a computer to determine whether investigators can assess mood and anxiety by analyzing speech and visual patterns. The audio and video will not be listened to nor watched by study personnel, only analyzed by a computer. The investigator's hope is that it will help others in the future by aiding in the assessment of psychological state. This study is being conducted at CMC ED only.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age 18 and over) who presents to the UHCMC ED voluntarily with no obvious psychological disturbance by self-report or nurse/provider initial assessment
* English-speaking
* Patients with non-emergent concerns of Emergency Severity Index (ESI) level 3, 4, or 5

Exclusion Criteria:

* Prisoners
* Patients who are deemed to be critically ill (including life or limb threatening illness) or unable to consent
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who score 5-9 on the PHQ-9 | Baseline
  Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring, and measuring severity of depression. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Percentage of participants who score 10-14 on the PHQ-9 | Baseline
  Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring, and measuring severity of depression. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Percentage of participants who score 15-19 on the PHQ-9 | Baseline
  Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring, and measuring severity of depression. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Percentage of participants who score 20-27 on the PHQ-9 | Baseline
  Patient Health Questionnaire (PHQ-9) is a multipurpose instrument for screening, diagnosing, monitoring, and measuring severity of depression. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Percentage of participants who score 5-9 on the GAD-7 | Baseline
  Generalized Anxiety Disorder (GAD-7) is a easy to preform initial screening tool for generalized anxiety disorder. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Percentage of participants who score 10-14 on the GAD-7 | Baseline
  Generalized Anxiety Disorder (GAD-7) is a easy to preform initial screening tool for generalized anxiety disorder. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Percentage of participants who score above 15 on the GAD-7 | Baseline
  Generalized Anxiety Disorder (GAD-7) is a easy to preform initial screening tool for generalized anxiety disorder. Questions are scored on a Likert scale of 0-3 with 0 being not at all and 3 being nearly every day.
Number of participants that AI screened positive for mild depression symptoms. | Baseline
Number of participants that AI screened positive for moderate depression symptoms. | Baseline
Number of participants that AI screened positive for moderately severe depression symptoms. | Baseline
Number of participants that AI screened positive for severe depression screening | Baseline
Number of participants that AI screened positive for mild anxiety symptoms. | Baseline
Number of participants that AI screened positive for moderate anxiety symptoms. | Baseline
Number of participants that AI screened positive for severe anxiety symptoms. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Faryar, MD, MPH, Principal Investigator — University Hospitals
Locations (1):
- University Hospitals ED, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No